**Title:** Diagnostic Accuracy of Artificial Intelligence, CBCT, and Clinical Examination in Detecting Number of Root Canals in Conventional and Retreated Maxillary and Mandibular Molars

NCT Number: "Pending"

**Date:** 29/10/2024

Informed consent Researcher's name:

determine

first

in

molars of

using 3D

the

detecting

accuracy

imaging.

the

the

to

the

program

methodand

Research Title: Diagnostic Accuracy of Artificial Intelligence, CBCT, and Clinical Examination in Detecting Number of Root Canals in Conventional and Retreated Maxillary and Mandibular Molars

| Patient's | | name: | | | | Age: | | Gender | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Addres | s: | | | | | | | | | | | |
| Phone: | | | | Mobile: | | | | | | | | |
| 1. Introduction: | | | We | ask | you | to | particij | oate | in | a | medica | ıl |
| researc | | eh | study. | Introdu | iction: | We | are | asking | you | to | partici | pate |
| | in | | medica | | | | study. | | docum | ent | contains | |
| | import | ant | inform | ation | about | the | reason | | the | study | and | what |
| | you | should | | if | you | choose | to | particij | pate | in | this | study. |
| | title<br>nation i<br>bular M | n Detec | | _ | | _ | | | _ | | | Clinical<br>lary and |
| 2. Participation | | | in | the | researc | h | is | volunta | arv | and | free | of |
| | charge | | are | no | burden | | or | costs | for | the | volunte | |
| | and | the | volunte | | has | the | right | to | withdra | | from | the |
| | research<br>voluntary<br>costs on | | at | any | time. | Partici | _ | in | the | researc | - | is |
| | | | and | free | of | charge | - | are | no | burden | | |
| | | | the | volunte | | and | the | volunte | | has | the | right |
| | | withdra | | from | the | researc | | at | any | time. | | 118114 |
| | | background | | and | purpose | | of | conducting | | the | research: | |
| | Dentists | | face | many | challen | | during | | canal | treatme | | |
| | includi | | the | failure | | detect | _ | canals | | the | root | canal |
| | system | _ | which | leads | to | incom | olete | disinfe | ction | and, | consea | uently, |
| | root | - | treatme | | | Scienti | | backgr | | and | researc | |
| | objecti | | Dentis | | face | | challen | _ | during | | canal | |
| | treatme | | includi | | the | failure | | detect | _ | the | canals | in |
| | the | root | | system | | which | | to | incomp | | disinfe | |
| | and | | uently | - | canal | failure | | aim | of | this | study | |

of

lower jaw

number

the

compared

artificial

root

to

of

intelligence

clinical

canals in

the

- 4. Research location: Clinics Complex, Faculty of Dentistry, Misr International University
- Research location: Clinic Complex, Facultyof Dentistry, Misr International University
- 5. Number of participants in the study: 212 patients Number of participants in the study: 212 patients
- 6.Method of selecting participants in the study:
- study selected from genders **Participants** in the are both aged 18-40 years, who adhere are interested in generaloral health, able to to follow-up conditions, do not suffer from any organicdisease. non-pregnant and non-lactating women, who do not regularly take painkillers antiinflammatory medications before the study date, and or history of allergy to of have no any the materials used in this study.
- 7. Details of the research steps: Details of the research steps:
- **Patients** who attend the dental clinics at the International University of Egypt and permanent molars requiring treatment have root canal criteria will or retreatment according to eligibility be selected. Informed consent will be obtained. and then two-dimensional before the X-rays will be conducted Three-dimensional treatment. imaging will performed for all cases. Other radiographs will be be avoided between treatments reduce the patient's to radiation. assigned exposure to **Patients** will be students specializing canal treatment. who will graduate in root procedure canals and then perform access the record to root a After comparing their number. the doctor's report with the 3D scans and artificial intelligence the program, the patient will be referred to the graduate students to complete the treatment procedures.
- 8. Duration of study: One patient within the trial. the day per Duration study: One patient within the of the day per trial.
- 9. Potential side effects of conducting the research: Potential side effects of conducting the research:
- The procedure may not be 100% successful, which could necessitate re-treatment or surgeryon the affected tooth.
- Pain may occur after the end of the root canal treatment session, swelling, inability or bruising, or to move several days the normally, which may last for jaw or more.

- Some tools may break inside the nerve during treatment, and thev can either be left as they are or surgically removed by a specialist.
- Some of the tools used may cause a hole in the tooth, which might require additional surgical intervention specialist by a tooth loss. could result in or
- Nerveinjury, which may temporary lead to and sometimes persistent numbness tingling the tongue, or other or in lips, chin, areas
- The tooth may need a post placement or filling reconstruction before the crown is placed.
- 10. benefits Expected of the research: reducing diagnostic failure. The errors that may lead root canal treatment to benefits research: diagnostic expected of the reducing canal treatment failure. errors that mav lead to root Secondly, reducing treatment time and increasing its accuracy, which will enhance treatment the successrate of your by eliminating human error.

information Confidentialityof your information: Your will be treated with confidentiality, researchers members complete and only and of ethics committee After the the will have access to your data. study is completed, will he informed results. you of the research You have the right answer any question you do not not to videos of wish to answer. Photographs or my teeth may solely for documentation, educational, be taken and used or focusing without showing research purposes, on the teeth the face.

11. Your right withdraw: You have the right withdraw to to from the research time without providing at any consequences for reasonsand without negative vou. Your any right to withdraw: You have the right to withdraw from the time without providing research at any reasonsand without negative consequences for you. any

In inquiries regarding case of any the treatment. a number will assigned for the research. be and you can contact it.

Name of the physician conducting the research: Salma Khaled Kamel (01000101236)

Position: Assistant Lecturer Misr International University I have reviewed acknowledge that I and understood the procedures that will be carried out through this research and agree to them. I

Participant in the research:

Name:

Signature (thumbprint):

First witness (if present/in case of verbal consent):

Date:

Researcher's signature:

Date: